CLINICAL TRIAL: NCT02233920
Title: Postmarketing Surveillance Study (as Per § 67(6) AMG [German Drug Law]) of Ventilat® Metered-dose Inhaler in Chronic Obstructive Bronchitis
Brief Title: Post-marketing Surveillance of Ventilat® Metered Dose Inhaler in Chronic Obstructive Bronchitis
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 54.564
Record Dates: First submitted 2014-09-08; First posted 2014-09-09 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Chronic obstructive bronchitis patients
  Interventions: Drug: Ventilat® - metered dose inhaler

INTERVENTIONS:
Drug: Ventilat® - metered dose inhaler

SUMMARY:
Study to obtain further information on the tolerability and efficacy of Ventilat® metered-dose inhaler in the treatment of Chronic Obstructive bronchitis under conditions of daily practice

ELIGIBILITY:
Inclusion Criteria:

* Primarily Patients of both genders older than 40 years, who suffer from Chronic Obstructive bronchitis
* Only patients who have not been treated with an anticholinergic within the last year are to be considered for inclusion

Exclusion Criteria:

•Contraindications listed in the Instructions for Use/Summary of Product Characteristics for Ventilat® metered dose inhaler

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with chronic obstructive bronchitis disease recruited at pneumologists
Sampling Method: Non-Probability Sample
Enrollment: 716 (Actual)
Dates: Start 2000-01; Primary Completion 2000-12 (Actual)

PRIMARY OUTCOMES:
Change in the clinical picture | after 4 weeks

SECONDARY OUTCOMES:
Assessment of efficacy by investigator on a 4-point scale | after 4 weeks
Assessment of efficacy by patient on a 4-point scale | after 4 weeks
Number of patients with adverse drug reactions | up to 4 weeks
Assessment of tolerability by investigator on a 4-point scale | after 4 weeks
Assessment of patient by investigator on a 4-point scale | after 4 weeks